CLINICAL TRIAL: NCT06238219
Title: Clinical Practice Survey on the Management of Neuromuscular Blocking Agents and Their Antagonism During General Anesthesia
Brief Title: Management of Neuromuscular Blocking Agents and Their Antagonism
Acronym: NMBA_periop
Status: Recruiting | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2024007
Record Dates: First submitted 2024-01-23; First posted 2024-02-02 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Neuromuscular Blocking Agents; Neuromuscular Monitoring
MeSH Terms: interventions — Neuromuscular Blocking Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NMBA cohort: Patients undergoing surgery under general anesthesia with use of neuromuscular blocking agents
  Interventions: Drug: Neuromuscular Blocking Agent

INTERVENTIONS:
Drug: Neuromuscular Blocking Agent — Administration of any neuromuscular blocking agent for surgery under general anesthesia

SUMMARY:
Neuromuscular blocking agents (NMBA) are commonly used in clinical practice during general anesthesia to facilitate induction, intubation and surgery. Some studies have shown that their use can be deleterious if not codified. Recent recommendations concerning their use and antagonization were published in 2023.

Research hypothesis:

Using a single-center, retrospective practice study, we aim to analyze whether the 2023 ASA and ESAIC recommendations are being implemented regarding the use of neuromuscular blocking agents.

ELIGIBILITY:
Inclusion Criteria:

- All patients undergoing surgery with use of neuromuscular blocking agents at our institution

Exclusion Criteria:

- Incomplete electronic anesthesia record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery with use of neuromuscular blocking agents at our institution from 2018 to 2023.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to ASA and ESAIC guidelines for the use and monitoring of neuromuscular bocking agents (%) | 10 hours
  Train of four (TOF) ratio and TOF-count, as well as post-tetanic count (PTC) will be extracted from the electronic anesthesia record together with the type, dosage and timing of neuromuscular blocking agents. At intubation, antagonisation and extubation, the use of monitoring, the correct dose for antagonising agents (neostigmine or sugammadex) will be recorded. Concordance with current guidelines from ASA (American society of anaesthesiologists) and ESAIC (European society of anaesthesia and intensive care) will be analysed with a Chi-square test (observed versus expected). The % of adherence to the guidelines will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire de Bruxelles - Hôpital erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirmeier E, Eriksson LI, Lewald H, Jonsson Fagerlund M, Hoeft A, Hollmann M, Meistelman C, Hunter JM, Ulm K, Blobner M; POPULAR Contributors. Post-anaesthesia pulmonary complications after use of muscle relaxants (POPULAR): a multicentre, prospective observational study. Lancet Respir Med. 2019 Feb;7(2):129-140. doi: 10.1016/S2213-2600(18)30294-7. Epub 2018 Sep 14. PMID 30224322
- [Background] Blobner M, Hunter JM, Meistelman C, Hoeft A, Hollmann MW, Kirmeier E, Lewald H, Ulm K. Use of a train-of-four ratio of 0.95 versus 0.9 for tracheal extubation: an exploratory analysis of POPULAR data. Br J Anaesth. 2020 Jan;124(1):63-72. doi: 10.1016/j.bja.2019.08.023. Epub 2019 Oct 10. PMID 31607388
- [Background] Fuchs-Buder T, Brull SJ. Is less really more? A critical appraisal of a POPULAR study reanalysis. Br J Anaesth. 2020 Jan;124(1):12-14. doi: 10.1016/j.bja.2019.09.038. Epub 2019 Nov 2. No abstract available. PMID 31685216
- [Background] Thilen SR, Weigel WA, Todd MM, Dutton RP, Lien CA, Grant SA, Szokol JW, Eriksson LI, Yaster M, Grant MD, Agarkar M, Marbella AM, Blanck JF, Domino KB. 2023 American Society of Anesthesiologists Practice Guidelines for Monitoring and Antagonism of Neuromuscular Blockade: A Report by the American Society of Anesthesiologists Task Force on Neuromuscular Blockade. Anesthesiology. 2023 Jan 1;138(1):13-41. doi: 10.1097/ALN.0000000000004379. PMID 36520073
- [Background] Fuchs-Buder T, Romero CS, Lewald H, Lamperti M, Afshari A, Hristovska AM, Schmartz D, Hinkelbein J, Longrois D, Popp M, de Boer HD, Sorbello M, Jankovic R, Kranke P. Peri-operative management of neuromuscular blockade: A guideline from the European Society of Anaesthesiology and Intensive Care. Eur J Anaesthesiol. 2023 Feb 1;40(2):82-94. doi: 10.1097/EJA.0000000000001769. Epub 2022 Nov 15. PMID 36377554